CLINICAL TRIAL: NCT04263805
Title: A Vignette-based Randomized Controlled Trial to Evaluate the Impact of Research Climate on Research Practices of Doctoral Students Facing Dilemma Situations
Brief Title: A Vignette-based Randomized Controlled Trial to Evaluate the Impact of Research Climate on Research Practices of Doctoral Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ISB-013
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: The Study Focus on no Specific Condition

STUDY DESIGN:
Masking Description: It is not possible to blind participants to the intervention. However, participants will be blinded to the study hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vignette with research climate (Experimental): Participants in this arm will receive vignettes describing a dilemma situation in research (e.g adding honorary author) with additional sentence describing research climate (i.e. an environment where their peer had detrimental practice in a similar situation)
  Interventions: Other: Vignette with emphasis on research climate
- Vignette without research climate (Active Comparator): Participants in this arm will receive vignettes describing a dilemma situation in research without the additional sentence describing research climate
  Interventions: Other: Vignette with emphasis on research climate

INTERVENTIONS:
Other: Vignette with emphasis on research climate — A vignette describing a dilemma situation for a researcher (e.g. adding an honorary author) with or without a research environment factor (i.e. an environment where other researchers commit detrimental research practice)

SUMMARY:
This study aims to evaluate the impact of research climate on PhD students' research practice (i.e., an environment where their peer (i.e., a post-doc researcher) had detrimental practice in a similar situation)

DETAILED DESCRIPTION:
PhD students are the next generation of researchers and will present the field in the future. However, several environmental factors might influence their research practice. In this study, the investigators will evaluate the impact of research climate on PhD students' research practice (exposure to an environment where their peers commit a detrimental practice).

Objective: To evaluate the impact of research climate on PhD students' research practice

Design: A randomized controlled trial

1. Intervention: Participants will be shown two case vignettes describing dilemma situations in research reported with and without research climate factor.
2. Participants: The participants will be PhD students in all biomedical disciplines.
3. Sample size will be 300 participants
4. Primary outcome: In each vignette, participants will have to indicate which solution they prefer on a semantic differential scale, rated from - 5 to -1 (preference for solution A) and from 1 to 5 (preference for solution B). Participants will be forced to make a choice between the 2 solutions. The primary outcome will be the mean preference score.
5. This study is approved by ethics review regulations by INSERM (CEEI-IRB): IRB00003888

ELIGIBILITY:
Inclusion Criteria:

* PhD students in biomedical disciplines

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
mean preference score | Immediate assessment
  In each vignette, participants will have to indicate which solution they prefer on a semantic differential scale, rated from - 5 to -1 (preference for solution A) and from 1 to 5 (preference for solution B).

SECONDARY OUTCOMES:
proportion of students who chose the detrimental research practice (DRP) | Immediate assessment
  Proportion of students rated from -5 to -1 for the DRP.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Epidémiologie Clinique, hôpital Hôtel Dieu, Assistance Publique-Hôpitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen VT, Sharp MK, Superchi C, Baron G, Glonti K, Blanco D, Olsen M, Vo Tat TT, Olarte Parra C, Neveol A, Hren D, Ravaud P, Boutron I. Biomedical doctoral students' research practices when facing dilemmas: two vignette-based randomized control trials. Sci Rep. 2023 Sep 29;13(1):16371. doi: 10.1038/s41598-023-42121-1. PMID 37773192